CLINICAL TRIAL: NCT00000292
Title: Acute Withdrawal From Smoked Cocaine
Brief Title: Acute Withdrawal From Smoked Cocaine - 9
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-9; P50-09259-9
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1996-04

CONDITIONS: Cocaine-Related Disorders; Substance Withdrawal Syndrome; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance Withdrawal Syndrome; Substance-Related Disorders | interventions — Cocaine

INTERVENTIONS:
Procedure: Cocaine

SUMMARY:
The purpose of this study is to develop an experimental paradigm to examine acute withdrawal symptoms from cocaine.

DETAILED DESCRIPTION:
Although there are clearly identifiable withdrawal syndromes following cessation of a number of abused drugs such as alcohol and heroin, it is unclear whether a withdrawal syndrome follows the cessation of crack cocaine. A laboratory model of withdrawal from smoked (crack) cocaine would provide a safe and systematic method of testing the efficacy of behavioral or pharmacological treatments for withdrawal symptoms following cocaine smoking cessation. Therefore, this study investigated acute behavioral, subjective, and physiological withdrawal symptomatology for 6 hrs following 7 deliveries of 2 dose sized (0.07 vs. 0.4 mg/kg) of smoked cocaine. The behavioral measure was performance on a computerized reaction time task, subjective measures included participant and observer ratings of mood and withdrawal symptomatology, and physiological measures comprised heart rate and blood pressure. It was hypothesized that signs and symptoms of withdrawal from smoked cocaine would be greater following the 0.4 mg/kg dose size, compared to the 0.07 mg/kg dose size.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-45 with a history of smoked cocaine use at least twice a week for the past six months, including 0.5 g of cocaine in a 24hr period on at least one occasion. In good health as evidenced by physical exam and complete blood count, chest X-ray and electrolyte and liver function tests, with a normal resting 12-lead electrocardiograph (ECG) and blood pressure of less than 140/90 mmHg. Using an acceptable method of birth control. Having a urine toxicology screen positive for cocaine metabolites.

Exclusion Criteria:

Any DSM-IV Axis I disorder other than cocaine abuse or dependence, or dependence or daily use of psychoactive drugs other than nicotine or caffeine. A history of violence and/or currently on probation, parole or awaiting trial. Pregnant as determined by serum pregnancy screen, lactating or having delivered a child in the past 12 months. Seropositive tests for the human immunodeficiency virus (HIV) or hepatitis B. History of seizure disorder.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-04; Study Completion 2001-12

PRIMARY OUTCOMES:
Behavioral
Subjective
Physiological measures

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States